CLINICAL TRIAL: NCT04566380
Title: A Multicenter, Open-label, Phase II Pan-Tumor Study in Patients Who Have Participated in Trials to Investigate Efficacy and Safety of ONO-4538 as Monotherapy or in Combination With Other Therapies and Are Continuing ONO-4538 Treatment (ONO-4538-98)
Brief Title: ONO-4538 Phase II Rollover Study (ONO-4538-98)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-98; jRCT2080225345 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Pan-tumor
MeSH Terms: interventions — Nivolumab; Oxaliplatin; S 1 (combination); Capecitabine; Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-4538 Monotherapy cohort (Experimental): 480 mg of ONO-4538 IV Q4W or 240 mg of ONO-4538 IV Q2W per the investigator's choice
  Interventions: Drug: ONO-4538
- Combination therapy cohort (Experimental): ONO-4538 at 360 mg IV Q3W or 480 mg IV Q4W, and Combination therapies (S-1 + Oxaliplatin [SOX] therapy , Capecitabine + Oxaliplatin [CapeOX] therapy , Bevacizumab or Temozolomide) selected by the principal investigator or subinvestigator in the Parent Study will be continued in this study.
  Interventions: Drug: ONO-4538; Drug: oxaliplatin; Drug: S-1; Drug: capecitabine; Drug: bevacizumab; Drug: temozolomide

INTERVENTIONS:
Drug: ONO-4538 — IV infusion over 30 minutes
Drug: oxaliplatin — IV infusion over 2 hours
  Arms: Combination therapy cohort
Drug: S-1 — Administered orally twice daily
  Arms: Combination therapy cohort
Drug: capecitabine — Administered orally twice daily
  Arms: Combination therapy cohort
Drug: bevacizumab — IV infusion over 30 minutes
  Arms: Combination therapy cohort
Drug: temozolomide — Administered orally once daily for 5 days every 28 days
  Arms: Combination therapy cohort

SUMMARY:
This study is intended to confirm the long-term safety of ONO-4538 in pan-tumor participants being treated with ONO-4538 monotherapy or in Combination with Other Therapies in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Participant who is being treated with ONO-4538 as monotherapy or in Combination with Other Therapies in clinical trials
2. Participant who is eligible for ONO-4538 monotherapy or in combination with other therapies as per the clinical trials, and/or investigator-assessed clinical benefit

Exclusion Criteria:

1. Participant judged to be incapable of providing consent for reasons such as concurrent dementia
2. Participant judged by the investigator to be inappropriate as participants of this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Aes) | From Day 1 up to 28 days after the end of the treatment phase
  (non)

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (38):
- Japan (22):
  - Chiba Clinical Site1, Kashiwa, Chiba
  - Ehime Clinical Site1, Matsuyama, Ehime
  - Fukuoka Clinical Site1, Kurume, Fukuoka
  - Hokkaido Clinical Site1, Sapporo, Hokkaido
  - Hyogo Clinical Site1, Akashi, Hyōgo
  - Kanagawa Clinical Site1, Yokohama, Kanagawa
  - Oita Clinical Site1, Yufu, Oita Prefecture
  - Osaka Clinical Site1, Suita, Osaka
  - Osaka Clinical Site3, Takatsuki, Osaka
  - Saitama Clinical Site1, Hidaka, Saitama
  - Saitama Clinical Site2, Kitaadachi-gun, Saitama
  - Tokyo Clinical Site3, Bunkyo-ku, Tokyo
  - Tokyo Clinical Site2, Chuo-ku, Tokyo
  - Tokyo Clinical Site1, Koto-ku, Tokyo
  - Tokyo Clinical Site4, Shinjuku-ku, Tokyo
  - Chiba Clinical Site2, Chiba
  - Fukuoka Clinical Site2, Fukuoka
  - Fukuoka Clinical Site3, Fukuoka
  - Hiroshima Clinical Site1, Hiroshima
  - Kyoto Clinical Site1, Kyoto
  - Okayama Clinical Site1, Okayama
  - Osaka Clinical Site2, Osaka
- South Korea (9):
  - Daegu Clinical Site1, Daegu
  - Gyeonggi-do Clinical site1, Gyeonggi-do
  - Incheon Clinical Site1, Incheon
  - Seoul Clinical Site1, Seoul
  - Seoul Clinical Site2, Seoul
  - Seoul Clinical Site3, Seoul
  - Seoul Clinical Site4, Seoul
  - Seoul Clinical Site5, Seoul
  - Seoul Clinical Site6, Seoul
- Taiwan (7):
  - Kaohsiung Clinical Site1, Kaohsiung City
  - Kaohsiung Clinical Site2, Kaohsiung City
  - Tainan Clinical Site1, Tainan
  - Tainan Clinical Site2, Tainan
  - Taipei Clinical Site1, Taipei
  - Taipei Clinical Site2, Taipei
  - Taoyuan Clinical Site1, Taoyuan District

IPD SHARING:
Plan to Share IPD: No